CLINICAL TRIAL: NCT05617235
Title: Investigation of The Effect of Kinesiology Tape on Pain, Respiratory Function and Respiratory Muscle Strength After Thoracotomy-A Randomized Controlled Study
Brief Title: Kinesiology Taping After Thoracotomy
Acronym: Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Neriman Temel Aksu, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Akdeniz Univ
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Post Operative Pain; Thoracotomy; Pulmonary Function
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy and Rehabilitation (No Intervention): A training will be given including information about the postoperative recovery process, the purpose of respiratory physiotherapy and rehabilitation, the importance of physiotherapy and rehabilitation in the postoperative period, attention to speed up recovery and prevention of complications, breathing exercises, coughing training, posture exercises, early mobilization and its importance, and answering patient questions.The program includes progressive ambulation and progressive shoulder and rib cage exercises. These exercises will be performed under the supervision of a physiotherapist from the first postoperative day. The exercises will be advanced every day by increasing the number of repetitions.
- Kinesiology taping (Experimental): On the postoperative 0th day, kinesiology taping was applied to the patients in the study group whose hemodynamic status was stable after extubation by an expert physiotherapist. All tapes were applied by the same physiotherapist on clean and shaved skin (if necessary). Investigators applied kinesiology taping as described below:
  1. In order to stimulate the facilitation of the diaphragmatic function, a 5 cm wide kinesiological tape was applied on the skin.
  2. Taping was applied to the latissimus dorsi and serratus anterior muscles, which were cut during the thoracotomy.
  3. In addition, kinesiology taping can be performed on the trigger pain point of the patient (usually above the pectoralis major).
  The kinesiology tape can stay for 3-4 days if the patient does not develop any discomfort. After 3-4 days, the tape was renewed. Thus, taping was done twice for each patient. The bands were removed at 1 week postoperatively.
  Interventions: Device: Kinesiology taping

INTERVENTIONS:
Device: Kinesiology taping — On the postoperative 0th day, kinesiology taping was applied to the patients in the study group whose hemodynamic status was stable after extubation by an expert physiotherapist. Investigators applied kinesiology taping as described below:
  1. In order to stimulate the facilitation of the diaphragmatic function
  2. Taping was applied to the latissimus dorsi and serratus anterior muscles, which were cut during the thoracotomy.
  3. In addition, kinesiology taping can be performed on the trigger pain point of the patient .
  After 3-4 days, the tape was renewed. Thus, taping was done twice for each patient. The bands were removed at 1 week postoperatively.
  Arms: Kinesiology taping

SUMMARY:
Effective pain control after thoracotomy increases the patient's respiratory functions and related quality of life, reduces the length of hospital stay and the amount of analgesia use. Kinesiology taping has been used in sports injuries for many years and has been used in recent years to reduce pain after major surgery. This study was conducted to examine the effect of kinesiology taping on pain, respiratory function and respiratory muscle strength in patients who underwent thoracotomy.In this prospective randomized controlled experimental study, individuals between the ages of 20-75 who underwent thoracotomy with posterolateral thoracotomy and who agreed to participate in the study were included. Unlike the control group, kinesiology taping was applied to the study group for 7 days after surgery. Pain, respiratory functions, respiratory muscle strength, amount of analgesic drug use, and quality of life were evaluated preoperatively, postoperative day 0, before tape application, postoperative 1st day, postoperative 2nd day, postoperative 7th day and postoperative 1st month.

DETAILED DESCRIPTION:
There are few studies showing the efficacy of kinesio taping for alleviating postoperative pain. Kinesio taping reduces postoperative pain, functional activity impairment, analgesic drug use, and lymphedema. Kinesio taping can improve cough reflex, secretion excretion, inspiratory muscle strength and respiratory function.Kinesio taping has been used in sports injuries for many years and has been used in recent years to reduce pain after major surgery. The aim of this study is to examine the effect of kinesio taping on pain, respiratory function and respiratory muscle strength after thoracotomy.This study was conducted on patients who underwent posterolateral thoracotomy. Written informed consent was obtained from each patient. The study protocol was approved by the Clinical Research Ethics Committee. The study was conducted in accordance with the principles of the Declaration of Helsinki. Patients were randomly assigned to 1:1 Kinesio taping group or control group using a computerized random number generator (GraphPad Software, San Diego, California) on postoperative day 0.The first group of the study consisted of patients in the Kinesio taping group, who underwent kinesio taping in addition to postoperative pulmonary rehabilitation and standard pain medication applications, and the second group consisted of patients in the control group, who underwent postoperative pulmonary rehabilitation and standard pain medication applications. On the postoperative 0th day, kinesiology taping was applied to the patients in the Kinesio taping group whose hemodynamic status was stable after extubation by an expert physiotherapist. The material we used for kinesio taping was Kinesio® Tex Gold™ (Kinesio Holding Corporation, Albuquerque, NM, USA), a 100% cotton, latex-free, 5 cm wide elastic band. A The kinesio tape can stay for 3-4 days if the patient does not develop any discomfort. After 3-4 days, the tape was renewed. The bands were removed at 1 week postoperatively.

The patients were followed from the preoperative period until discharge. For each patient, age, gender, weight and height measurements, educational status, type of surgery, whether there is any additional systemic disease, smoking, alcohol habits, medications they constantly use, previous operations, postoperative complications, surgical procedure, duration of operation, duration of anesthesia, Chest tube incision time and hospital stay were recorded.

The G*power sample size calculator was used to determine the sample size of the study. A sample size of 35 subjects for each group was estimated, assuming sample size, 0.05 type I error rate (α) and 90% power (1-α). A total of 88 patients were included to avoid possible loss or exclusion. Statistical analysis was performed using the SPSS version 23 statistical software program (SPSS Inc., Chicago, IL). In the comparisons between the two groups, Student's t test or Mann-Whitney U test was used. Chi-square test (Fisher exact test, 2-tailed) was used to compare categorical variables. Two-way analysis of variance was used in repeated measures to evaluate the change over time of the measured variables of the treatment and control groups and the group-time interactions.

ELIGIBILITY:
Inclusion Criteria:

* Who underwent thoracotomy with a posterolateral thoracotomy incision
* Who agreed to participate in the study, were aged 20-75 years
* Who had no known cerebrovascular disease
* Who had no morbid obesity and heart disease that would interfere with the study
* Who had no cognitive and cognitive impairments that would interfere with communication

Exclusion Criteria:

* Who had chest trauma, thoracotomy or tube thoracostomy
* Who had not complying with the pulmonary function test
* Who are allergic to the tape

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change of Pain Score | Change from Baseline Pain Score at 4 weeks.
  The Visual Analog Scale (VAS) was used as a one-dimensional scale for pain assessment. VAS is a self-administered, one-dimensional measure of pain intensity widely used in various adult populations. The VAS is a 10 cm long line in which participants mark the point they believe best represents the severity of pain. Always "0" means no pain, while "10" means excruciating pain.
  When asked, patients touch a point corresponding to their degree of pain, and this mark indicates the degree of pain on the scale. Higher scores indicate greater pain severity. Preoperative, postoperative day 0, pre-taping, postoperative 1st day, postoperative 2nd day, postoperative 7th day and postoperative 1st month were evaluated.
Change of Pulmonary Function | Change from Baseline Pulmonary Function at 4 weeks.
  Pulmonary function testing was performed using a digital spirometer (Pony FX, COSMED Inc., Italy) with subjects in a comfortable 90-degree sitting position.This test was repeated 3 times for each patient and the best value was recorded. A 1-minute rest period was given between each test. Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), 1 second forced expiratory volume to forced vital capacity (FEV1/FVC), peak expiratory flow (PEF), 25-75% forced expiratory flow (FEF25-75) have been recorded. The tests were performed preoperatively, postoperative day 0, before tape application, postoperative day 1, postoperative day 2, postoperative day 7, and postoperative 1 month.
Change of Respiratory Muscle Strength | Change from Baseline Pulmonary Strenght at 4 weeks.
  Respiratory muscle strength was evaluated by measuring maximal inspiratory and maximal expiratory pressures with a portable intraoral pressure measuring device (Pony FX, COSMED Inc., Italy). During the measurements, participants were verbally encouraged for maximum performance. The maneuvers were repeated at least 5 times at intervals of at least 30 seconds, and the best among the measurements with a 5-10% difference was selected for analysis. MIP and MEP values were determined as cmH2O. The tests were performed preoperatively, postoperative day 0, before tape application, postoperative day 1, postoperative day 2, postoperative day 7, and postoperative 1 month.
Change of Quality of Life | Change from Baseline Quality of Life at 4 weeks.
  The Short Form-36 (SF-36) quality of life scoring was used to evaluate the quality of life of the patients. SF-36 is a questionnaire with 8 subscales that gives information about the health status and quality of life of the person. SF-36 was translated into Turkish in 1999. Confirmation studies were conducted in different patient groups.The tests were applied in the preoperative period, at the postoperative 1st month.

SECONDARY OUTCOMES:
Height in Meters | Initial assessment before surgery
  The height of all subjects in meters (m) will be noted before the surgery.
Weight in Kilograms | Initial assessment before surgery
  The weight of all subjects in kilograms (kg) will be noted before the surgery.
Body Mass Index (BMI) in kg/m^2 | Initial assessment before surgery.
  Body Mass Index (BMI) will be calculated with the formula weight (kg)/height (m)^2.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman Temel Aksu, Principal Investigator — Akdeniz Üniversitesi Antalya Sağlık Yüksekokulu
Locations (1):
- Neriman Temel Aksu, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No